CLINICAL TRIAL: NCT06693934
Title: Jockey Club Precision Prevention Programme on Young Onset Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Juliana CN Chan (Other)
Collaborators: Chinese University of Hong Kong (Other); St. James' Settlement (Other); Asia Diabetes Foundation (Other)
Responsible Party: Sponsor-Investigator, Juliana CN Chan, Professor, Asia Diabetes Foundation
Organization: Asia Diabetes Foundation (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRE-2024.243
Record Dates: First submitted 2024-10-28; First posted 2024-11-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Pre Diabetes; Hypertension; Dyslipidemia; Obesity
Keywords: Diabetes; Pre Diabetes; YOD; DM; Young Onset diabetes; Genetic test; Management; Prevention; Hypertension; Dyslipidemia; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Hypertension; Dyslipidemias; Obesity | interventions — Risk Assessment; Glucose Tolerance Test; Dosage Forms; Continuous Glucose Monitoring; Physical Examination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low risk (Other): Low risk progressors are those who are in the bottom 75% of the risk score based on both clinical and biogenetic risk markers
  Interventions: Genetic: Risk assessment with biogenetic and clinical test to predict diabetes risk; Behavioral: Education webinars, workshops and health messages
- High risk progressors (Other): High risk progressors are those who are in the top 25% of the risk score based on both clinical and biogenetic risk markers. They will undergo yearly OGTT to detect undiagnosed diabetes or impaired glucose tolerance (IGT) for early intervention. They will also receive low intensity team-based care with regular empowerment using webinars and whatsapp messages for 2 years.
  Interventions: Genetic: Risk assessment with biogenetic and clinical test to predict diabetes risk; Diagnostic Test: Oral glucose tolerance test (OGTT) and cardiovascular-kidney-metabolic (CKM) risk factors; Drug: Medication; Device: Continuous glucose monitoring (CGM) devices and/or weighing scale; Behavioral: Visit to family doctor with nurse education; Behavioral: Education webinars, workshops and health messages
- Impaired glucose tolerance (IGT) (Other): Subjects with IGT will receive team-based care including lifestyle modification and early use of metformin, subsidized weighing scale and CGM, supplemented by WhatsApp messages and webinars for empowerment for 2 years
  Interventions: Genetic: Risk assessment with biogenetic and clinical test to predict diabetes risk; Diagnostic Test: Oral glucose tolerance test (OGTT) and cardiovascular-kidney-metabolic (CKM) risk factors; Drug: Medication; Device: Continuous glucose monitoring (CGM) devices and/or weighing scale; Behavioral: Visit to family doctor with nurse education; Behavioral: Education webinars, workshops and health messages
- Diabetes (Other): Subjects with newly diagnosed diabetes will receive team-based care with structured assessment, JADE personalized report, testing for autoimmune markers, , subsidized CGM, weighing scale and medications with regular WhatsApp messages and webinars for empowerment for 2 years
  Interventions: Genetic: Risk assessment with biogenetic and clinical test to predict diabetes risk; Diagnostic Test: Oral glucose tolerance test (OGTT) and cardiovascular-kidney-metabolic (CKM) risk factors; Drug: Medication; Device: Continuous glucose monitoring (CGM) devices and/or weighing scale; Behavioral: Visit to family doctor with nurse education; Diagnostic Test: Joint Asia Diabetes Evaluation (JADE) assessment; Behavioral: Education webinars, workshops and health messages

INTERVENTIONS:
Genetic: Risk assessment with biogenetic and clinical test to predict diabetes risk — All participants will undergo genetic test and clinical measurement including body weight, body height, blood pressure, waist circumference and capillary blood glucose to predict diabetes risk with report explanation by doctors (for high risk, IGT and DM) and nurses (low risk). Genetic report will be updated annually for high risk and IGT group using updated clinical factors (e.g. age, BMI, BP).
Diagnostic Test: Oral glucose tolerance test (OGTT) and cardiovascular-kidney-metabolic (CKM) risk factors — High risk progressors will undergo OGTT and measurement of CKM factors at baseline. In those without IGT or diabetes, they will undergo OGTT and CKM risk factor assessment annually for 2 years. The IGT group will additionally have measurement of beta-cell function (HOMA indexes) and the DM group will additionally have autoimmune marker measurement.
  Arms: Diabetes; High risk progressors; Impaired glucose tolerance (IGT)
Drug: Medication — Nurse and medical consultations and subsidized medications (metformin, statin, ARB) will be provided to the high risk progressor, IGT and diabetes groups as appropriate for control of glucose and CKM risk factors.
  Arms: Diabetes; High risk progressors; Impaired glucose tolerance (IGT)
Device: Continuous glucose monitoring (CGM) devices and/or weighing scale — All high risk progressors will be given subsidized weighing scale and low-intensity laboratory assessments, nurse and doctor consultation, regular WhatsApp messages and webinars for 2 years. The IGT and DM group will receive additional subsidized CGM devices for empowerment.
  Arms: Diabetes; High risk progressors; Impaired glucose tolerance (IGT)
Behavioral: Visit to family doctor with nurse education — All participants in high risk, IGT and diabetes groups will have regular follow-up by family doctors and nurses.
  Arms: Diabetes; High risk progressors; Impaired glucose tolerance (IGT)
Diagnostic Test: Joint Asia Diabetes Evaluation (JADE) assessment — Participants found to have diabetes on OGTT will undergo annual JADE assessment which include eye/foot/urine/blood tests with issue of a personalized JADE report. The JADE Program is a quality improvement program to improve self management and inform shared decision making between doctor and patient.
  Arms: Diabetes
Behavioral: Education webinars, workshops and health messages — All participants would join the webinars. High risk progressors, IGT and DM group will receive regular WhatsApp messages, webinars and workshops.

SUMMARY:
This is a community-based implementation program consisting of multiple components delivered by a multidisciplinary team to detect and prevent young onset diabetes with precision and value using biogenetic markers, digital tools, integrated care through public private partnership. Adults aged between 18 and 44 (inclusive) without known diabetes and with at least one risk factor for diabetes will undergo a saliva DNA and capillary blood test and complete a questionnaire. Depending on their risk levels, participants will be stratified to high risk and low risk progressors to diabetes. The high risk progressors will undergo annual oral glucose tolerance test to detect diabetes and impaired glucose tolerance (IGT). All participants will receive a personalized report indicating their genetic and modifiable risk explained by nurses or doctors. All participants will be offered regular access to webinars for education and empowerment for 2 years. The high risk group will additionally receive a 2-year risk-stratified intervention with different combinations of care interventions. These include clinical and laboratory assessment for comprehensive evaluation of cardiovascular-kidney-metabolic risks, medical and nurse consultations, empowerment by health messages, webinars, face-to-face workshops, subsidies for medications and self-monitoring tools (e.g. CGM devices, weighing scale) to motivate behavioural change. The outcomes will be analysed within the REAIM framework (reach, effectiveness, adoption, implementation and maintenance), progresssion to prediabetes or diabetes, patient reported outcomes and cost effectiveness.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

In Hong Kong, 1 in 10 adults have diabetes. In hospital-based clinic setting, 1 in 5 adults with diabetes were diagnosed before the age of 40, i.e. young-onset diabetes (YOD). The latter is the major driver of recurrent hospitalizations, critical illnesses and premature death. Compared to fasting plasma glucose (FPG) or HbA1c, 2-hour PG is needed to detect impaired glucose tolerance (IGT) and diabetes (DM). Besides, 2-h PG is more robust than FPG or HbA1c in predicting major events and death. The selection of participants with IGT for intervention is based on the positive effects of lifestyle modification and metformin only in individuals with IGT and not in individuals with isolated IFG in randomized clinical trials. Besides, there is strong familial tendency of YOD and based on our published and in-house 20-year prospective data in a workforce, 80% of people who developed DM came from 20-30% of individuals with high genetic risk unmasked by modifiable risk factors such as obesity and smoking.

In this implementation project, investigators shall use a 2-stepped approach to identify adults aged between 18 and 44 (inclusive) with genetic predisposition to undergo yearly OGTT to diagnose IGT and diabetes early for intervention. Investigators shall apply the proprietary DForesee (DF) risk algorithm including clinical and biogenetic risk factors to select the top 25% of participants at the highest risk for IGT or diabetes in next 10 years to undergo yearly OGTT accompanied by a risk-based intervention program.

STUDY DESIGN AND METHODS:

By using quasi-experimental design based on an evidence-based multi-component strategy, investigators aim to detect and delay the onset of diabetes in adults aged less than 45 years. Investigators aim to identify 9,000 adults aged between 18 and 44 years (inclusive) in community- and clinic settings during a 2-year period, followed by 2 years of risk-stratified intervention. Investigators shall use clinical and biogenetic assessment including DNA testing, capillary blood test and administration of questionnaires to classify participants to high risk and low risk progressors. All participants will receive risk-based intervention. Low risk progressors will receive a personalized report indicating their genetic and modifiable risk explained by nurses and with repeated clinical and biogenetic assessment at year 2. The high risk progressors will additionally undergo annual oral glucose tolerance test to detect diabetes and impaired glucose tolerance (IGT) and will receive a personalized report explained by doctors. All participants will be offered regular access to webinars for education and empowerment for 2 years. The high risk group will additionally receive a 2-year risk-stratified intervention with different combinations of care interventions. These include clinical and laboratory assessment for comprehensive evaluation of cardiovascular-kidney-metabolic risks, medical and nurse consultations, empowerment by health messages, webinars, face-to-face workshops, subsidies for medications and self-monitoring tools (e.g. CGM devices for IGT and DM groups only, weighing scale for all high risk progressors) to motivate behavioural change.

INCLUSION and EXCLUSION CRITERIA Age 18-44 (inclusive) years without known diabetes, at least one risk factor for diabetes and with usual place of residence in Hong Kong, The risk factors for diabetes include central or general obesity, family history of diabetes, smoking history, history of hypertension, high blood glucose level, abnormal lipid level/ vascular disease, or fatty liver, history of gestational diabetes polycystic ovary syndrome or delivery of baby≥ 4kg (for women only), less than 150mins of physical activity every week.

People with known diabetes or conditions considered to be unsuitable by the project team including illiteracy will be excluded.

OUTCOME MEASURES The outcomes will be analysed within the REAIM framework (reach, effectiveness, adoption, implementation and maintenance), progresssion to prediabetes or diabetes, patient reported outcomes and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 44 years old
* With at least one risk factor for diabetes

Exclusion Criteria:

* Known history of Diabetes
* With conditions considered not suitable by the project team (including illiteracy)

The risk factors for diabetes include central or general obesity, family history of diabetes, smoking history, history of hypertension/ high blood glucose level/ abnormal lipid level/ vascular disease/ fatty liver, history of gestational diabetes/ polycystic ovary syndrome/ delivery of baby≥ 4kg (for women only), and less than 150mins of physical activity every week.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9000 (Estimated)
Dates: Start 2024-11-23 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of prediabetes or diabetes in the high and low risk progressor groups | From the date of recruitment until the end of the programme in 2 years.
  DForesee risk score will be used to define the high and low risk progressor groups at baseline and oral glucose tolerance test (OGTT) will be used to detect IGT or diabetes in the high risk progressor group and 10% of low risk progressor group.
  DForesee risk score consists of the overall risk for prediabetes and the overall risk for type 2 diabetes which will have 4 different risk levels including low, moderate, high and very high risk.

SECONDARY OUTCOMES:
The conversion rate of glycaemic status including Impaired fasting glucose (IFG), Impaired glucose tolerance (IGT) and diabetes over the study period | From the date of recruitment until the end of the programme in 2 years.
  The conversion rate of impaired fasting glucose (IFG), impaired glucose tolerance (IGT) and diabetes will be assessed for all high risk progressors using OGTT at baseline and annually. In addition,1 in 10 of the low risk progressors will also undergo OGTT at baseline and year 2 to ascertain their conversion rate to IGT or diabetes.
Change in the HbA1c over the study period | From the date of recruitment until the end of the Programme in 2 years
  High risk progressors will undergo yearly assessment to evaluate the HbA1c to determine the change in the blood glucose level during the program periods.
Change in the blood glucose level including FPG and 2-hour PG over the study period | From the date of recruitment until the end of the Programme in 2 years
  High risk progressors will undergo yearly assessment to evaluate the blood glucose level including FPG and 2-hour PG to determine the change in the blood glucose level during the program periods. In addition, 1 in 10 of the low risk progressors will evaluate the blood glucose level including FPG and 2-hour PG at baseline and year 2.
Change in the blood pressure level over the study period | From the date of the recruitment until the end of the Programme in 2 years
  High risk progressors will measure the blood pressure including the systolic and diastolic blood pressure at least once a year to evaluate the change or control of blood pressure. In addition, low risk progressors will also measure the blood pressure at baseline and year 2.
Change in lipids level including total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides over study period | From the date of recruitment until the end of the programme in 2 years
  High risk progressors will undergo yearly assessment to evaluate the control and changes of lipids throughout the study period.
Change in body weight over the study period | From the date of the recruitment until the end of the programme in 2 years
  High risk progressors will undergo yearly assessment to evaluate the change in body weight over the study period. Low risk progressors will also measure the body weight at baseline and year 2.
Change in waist circumference over the study period | From the date of the recruitment until the end of the Programme in 2 years
  High risk progressors will undergo yearly assessment to evaluate the change or control of waist circumference. Low risk progressors will also measure the waist circumference at baseline and year 2.
Change in albuminuria over the study period | From the date of the recruitment until the end of the programme in 2 years
  High risk progressors will undergo yearly assessment to evaluate the change in albuminuria over the study period.
Change in health literacy over the study period by using questionnaire | From the date of recruitment until the end of the programme in 2 years
  Questionnaire will be used by all participants to assess the health literacy by comparing the number of questions being answered correctly at baseline and at year 2 of the programme. The questionnaire consists of 10 multiple choice questions with 5 options including the questions about the health knowledge on 4 highs (diabetes, hypertension, dyslipidemia and obesity) and healthy diet. There will be one point for each question with a total of 10 points. The higher scores mean a better outcome.
Quality of life using EuroQoL with 5 demensions and 3 levels (EQ-5D-3L) Questionnaire | From the date of recruitment until the end of the programme in 2 years
  Questionnaire will be used to assess the quality of life (EuroQoL - EQ-5D-3L) of all participants at baseline and year 2. The EQ-5D-3L essentially consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three levels: no problems, some problems, and extreme problems (labelled 1-3).
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale numbered from 0 to 100. The endpoints are labelled 'The best health you can image' at number 100 and 'The worst health you can image' at number 0. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Change in lifestyles including eating habits, exercises, sleeping habits, smoking and alcohol over the study period by using questionnaire | From the date of recruitment until the end of the programme in 2 years
  Questionnaire, adopted from the questionnaire of a health promotion campaign named "Better Health for a Better Hong Kong", will be used to assess the change in lifestyles of all participants including eating habits, exercises, sleeping habits, smoking and alcohol at baseline and year 2.
  The questionnaire consists of 38 questions with multiple choice and free text questions which will enquiry about the intake frequency and serving of different food types, frequency, duration and intensity of exercises, smoking and drinking frequency, sleeping duration, etc.
The number of usage in healthcare resources such as clinic visits and hospital admissions | From the date of recruitment until the end of the programme in 2 years
  The number of usage in healthcare resources such as clinic visits and hospital admissions by self reporting by the participants during nurse and doctor consultations of high risk progressors and information from publicly available resources for all participants.
Cost-effectiveness analysis by mearsuring the transition rate of progression from normal glucose tolerace to IGT and IGT to diabetes during 4 year programme | From the date of recruitment until the end of the programme in 2 years
  A Markov model will be developed to evaluate the cost-effectiveness of the study by measuring the transition rate of progression from normal glucose tolerance to IGT and IGT to diabetes during the programme period. Cost effectiveness results will be estimated using incremental cost effectiveness ratios (ICER) derived by dividng the difference in total costs by difference in health outcome or effect (QALYs or YLL).

CONTACTS AND LOCATIONS:
Overall Officials: Juliana CN Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Asia Diabetes Foundation, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Consent for sharing of individual data have not been sought from participants. Summary statistics may be shared depending on nature of request